CLINICAL TRIAL: NCT06226077
Title: Project SHINE (Sleep Health INitiative for Equity): Culturally Informing a Sleep Extension Intervention for African American Adults
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022LS170 (B)
Record Dates: First submitted 2024-01-16; First posted 2024-01-26 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Insufficient Sleep
MeSH Terms: conditions — Obesity; Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: The intervention is a 6-week (4-week intervention, 1- week pre/post actigraphy measurement) 2-armed randomized control trial with the sleep extension intervention in one arm, and then an education contact control in the second arm.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sleep extension intervention arm (Experimental): sedentary and short sleep (=<6 hrs/night) African American adults with overweight/obesity randomized to the sleep extension intervention.
  Interventions: Behavioral: sleep extension intervention
- education contact control arm (Active Comparator): sedentary and short sleep (=<6 hrs/night) African American adults with overweight/obesity randomized to contact control intervention.
  Interventions: Behavioral: contact control intervention

INTERVENTIONS:
Behavioral: sleep extension intervention — The sleep intervention aims to increase sleep duration by one-hour (15 minutes/week) over the course of 4-weeks using components from Cognitive Behavioral Therapy for Insomnia. More specifically, the intervention consists of psychoeducation, sleep extension, sleep hygiene, and stimulus control. Participants will meet with Dr. Wu or a trained staff member once a week over the course of 4-weeks via Zoom. The intervention will be adapted based on feedback from the community, knowledge gained during previous interviews.
  Arms: sleep extension intervention arm
Behavioral: contact control intervention — The control condition is a contact-control intervention whereby participants will meet with Dr. Wu or a trained staff member once-week over the course of 4-weeks to receive education materials from the Healthy Homes intervention developed by the UT School of Public Health.
  Arms: education contact control arm

SUMMARY:
The proposed research aims to reduce obesity-related health disparities by promoting healthy lifestyle behaviors among African Americans (AAs), given the high disease burdens associated with low physical activity, insufficient sleep, and obesity. There will be two phases to the proposed research. Phase 1 (Aim 1) will encompass formative research and community engagement activities, and Phase 2 (Aim 2a and 2b) will be a randomized clinical trial.

The primary goal of Aim 1 is to conduct in-depth qualitative interviews in order to: (1) better understand sleep-related social contextual factors, knowledge, behaviors, and beliefs, and (2) discuss and receive feedback on an existing sleep intervention design and materials. The primary goal of Aim 2 is to explore the feasibility, satisfaction, and preliminary efficacy of a sleep intervention to increase sleep and physical activity (PA) among sedentary and short sleeping (≤6 hrs/night) African American adults with overweight/obesity, compared to a contact control group. (Aim 2a) An additional exploratory (Aim 2b) examines changes in cancer-relevant biomarkers between those who received the intervention vs the control condition (n = 20). Data will be collected from a sample of 20 participants (10 per condition) who volunteer to have their blood drawn pre- and post-intervention.

There are two phases of the study, and information gained during Phase 1 (Aim 1) will be used to inform Phase 2 (Aim 2). Thus, additional modifications to the protocol will be submitted prior to engagement in Phase 2.

ELIGIBILITY:
Inclusion Criteria:

Phase 1:

* Not meeting Physical Activity Guidelines
* age range: 21 to 75 years
* body mass index: ≥25.0 kg/m2
* average self-reported habitual sleep duration of ≤6 hours
* self-identify as Black or African American

Phase 2:

* Not meeting Physical Activity Guidelines
* age range: 21 to 75 years
* body mass index: ≥25.0 kg/m2
* average self-reported habitual sleep duration of ≤6 hours
* self-identify as Black or African American

Exclusion Criteria:

Phase 1:

* Self-reported organ-related disorder (COPD, cardiac arrhythmia, gastro-esophageal disorder)
* pregnant or less than 4 months postpartum
* infant living in household less than 1 year old

Phase 2:

* Self-reported organ-related disorder (COPD, cardiac arrhythmia, gastro-esophageal disorder)
* pregnant or less than 4 months postpartum
* infant living in household less than 1 year old

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the sleep intervention | 10 weeks
  feasibility is defined as 75% intervention attendance (3/4 sessions)
Satisfaction with the sleep intervention | 10 weeks
  satisfaction is defined as Client Satisfaction Questionaire score >=20, range 8-32, with higher scores indicating higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Wu, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States